CLINICAL TRIAL: NCT02030561
Title: Phase I/II Study of Expanded, Activated Autologous Natural Killer Cell Infusions With Trastuzumab for Patients With HER2+ Breast and Gastric Cancer
Brief Title: NK Cell Infusions With Trastuzumab for Patients With HER2+ Breast and Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC01/21/13; 2013/00566 (Other: Singapore NHG Domain Specific Review Boards)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer; Gastric Cancer
Keywords: NK cells; trastuzumab; immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab + NK cells (Experimental): During cycle 1, Day 1 patient will receive intravenous trastuzumab and subcutaneous IL-2 on day 1, followed by NK cell infusion on day 2, followed by subcutaneous IL-2 for an additional 5 doses three times a week to support NK cell viability and expansion in vivo.
  From cycles 2-4, patient will receive trastuzumab monotherapy alone every 21 days, except for patients who achieve objective tumor response after 2 cycles of therapy, who will then receive an additional infusion of NK cells along with trastuzumab during cycle 4 therapy at the same dose and schedule as in cycle 1.
  Patients will be taken off study after cycle 4, unless the patient has objective tumor response after 4 cycles of therapy with only stable disease after cycle 2, in which case the patient will be given another 2 cycles of trastuzumab with an additional NK cell infusion during cycle 6 therapy at the same dose and schedule as in cycle 1.
  Interventions: Drug: Trastuzumab + NK cells

INTERVENTIONS:
Drug: Trastuzumab + NK cells
  Other Names: Herceptin

SUMMARY:
This study will determine the safety and efficacy of expanded activated autologous NK cells administered after Trastuzumab in patients with HER2-positive breast or gastric cancer. It will also provide valuable insights of the role of NK cell infusions in adult solid tumors.

DETAILED DESCRIPTION:
Recently, targeted immunotherapies have become part of the therapeutic arsenal in adult solid tumors, and have shown promising activity in melanomas and prostate cancers. Trastuzumab is a monoclonal antibody that targets HER2 and is used routinely in combination with chemotherapy in HER2 over-expressing breast and gastric cancer. Trastuzumab is known to induce antibody dependent cell cytotoxicity (ADCC), among its various mechanisms for tumor cell kill. As such, trastuzumab may suitably be combined with immunotherapy as a strategy to harness the host's immune system against HER2-positive tumor cells.There is mounting evidence that natural killer (NK) cells have powerful anti-cancer activity. In patients with leukemia undergoing allogeneic hematopoietic stem cell transplant, several studies have demonstrated NK-mediated anti-leukemic activity. Allogeneic NK cell infusions in patients with primary refractory or multiple-relapsed leukemia have been shown to be well tolerated and void of graft-versus-host disease (GVHD) effects. In this study, we seek to enhance the antitumor activity of a commonly used antibody to treat HER2+ breast and gastric cancer, trastuzumab, administered in combination with infusion of activated and expanded autologous NK cells.This is a lead-in phase I followed by a phase II study. Up to 9 patients will be enrolled in phase I to test two different doses of NK cells to be infused into the patient. This will then be followed by a phase II study where 20 patients will be enrolled. Eligible patients will undergo apheresis about 9 days (up to 11 days) prior to cycle 1 therapy to harvest NK cells. The collected NK cells will be expanded and activated ex vivo. On day 1 of cycle 1, the patient will receive herceptin and subcutaneous IL2, followed by NK cell infusion on day 2 of cycle 1. This will then be followed by 5 doses of s/c IL2 three times a week to keep the NK cells activated in vivo. The patient will then receive three more cycles of herceptin (every 21 days). In patients who achieve objective tumor response after cycle 2 or cycle 4, a second NK cell infusion along with s/c IL2 will be administered with cycle 4 or cycle 6 herceptin respectively.This study will determine the safety and efficacy of this novel therapeutic strategy in HER2 positive breast and gastric cancer. It will also provide valuable insights of the role of NK cell infusions in adult solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Histologically confirmed diagnosis of HER2-positive breast or gastric cancer (defined as IHC 3+ or HER2 FISH amplification ratio >2.2)
3. Metastatic disease
4. Presence of measurable tumour by RECIST 1.1 criteria
5. Must have failed at least two lines of trastuzumab-containing systemic therapy (documented relapse while receiving adjuvant or neoadjuvant trastuzumab for HER2 positive breast cancer is eligible)
6. At least two weeks since receipt of any biological therapy, chemotherapy, and/or radiation therapy
7. Left ventricular ejection fraction ≥50%
8. Adequate organ function ANC ≥ 1500/µL Platelet count ≥ 100,000/µL Creatinine clearance ≥60ml/minute Total bilirubin ≤ 1.5 x upper limit normal (ULN) AST ≤ 2 x upper limit normal ALT ≤ 2 x upper limit normal
9. ECOG performance status of 0-1
10. Life expectancy of at least 60 days
11. Negative serum or urine pregnancy test result within 14 days prior to enrolment for women who are of childbearing potential
12. Ability to provide informed consent. Otherwise, a legally authorized representative (LAR) must be present throughout the consent process and is allowed to give consent on the patient's behalf.
13. Patients with reproductive potential must agree to use an approved contraceptive method
14. Ability to comply with study procedures

Exclusion Criteria:

1. Treatment within the last 30 days with any investigational drug
2. Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy
3. Major surgery within 28 days of study drug administration
4. Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
5. Lactating or pregnant.
6. Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator; serious cardiac illness or medical conditions including but not limited to:

   * Patients with dyspnea at rest.
   * History of documented congestive heart failure
   * High risk uncontrolled arrhythmias
   * Angina pectoris requiring a medicinal product
   * Clinically significant valvular disease
   * Evidence of transmural infarction on ECG
   * Poorly controlled hypertension
7. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment
8. Symptomatic brain metastases
9. Receipt of steroids during time period of 3 days prior to expanded NK cell infusion to 30 days after infusion (i.e. day -3 to day +30).

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 12-18 weeks
  During cycle 1 (21 days) and for at least 21 days following a second NK cell infusion if administered:
  - Patients will be reviewed twice a week with
  * Limited physical examination to include blood pressure, heart rate, weight
  * Full blood count, renal function and liver function tests
  * Toxicity rating using the NCI CTC scale
  * Concomitant medication notation and number of units required for transfusions
  Any significant abnormalities or significant toxicities have to be followed until recovery to baseline or 30 days after patient withdraws from the study, whichever occurs later.
  During other cycles when only trastuzumab is administered (without NK cells infusion or IL-2) Patients will be reviewed once every cycle of every 3-weekly cycle
Duration of Tumor Response Measure | Up to 36 months
  Among tumor responders, the duration of tumor response is measured from the date of enrolment until the first date of documented disease progression or death due to any cause, whichever occurs first. Duration of tumor response will be censored at the date of the last follow-up visit for tumor responders who are still alive and who have not progressed.
Time-to-Event Outcome Measure | Up to 36 months
  Time to documented disease progression is defined as the time from the date of enrolment to the first date of documented disease progression. Time to documented disease progression will be censored at the date of death for patients who have not had documented disease progression. For patients who are still alive at the time of analysis and who have not had documented disease progression, time to documented disease progression will be censored at the date of the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - National University Hospital, Singapore

REFERENCES:
- [Background] Beano A, Signorino E, Evangelista A, Brusa D, Mistrangelo M, Polimeni MA, Spadi R, Donadio M, Ciuffreda L, Matera L. Correlation between NK function and response to trastuzumab in metastatic breast cancer patients. J Transl Med. 2008 May 16;6:25. doi: 10.1186/1479-5876-6-25. PMID 18485193
- [Background] Voskens CJ, Watanabe R, Rollins S, Campana D, Hasumi K, Mann DL. Ex-vivo expanded human NK cells express activating receptors that mediate cytotoxicity of allogeneic and autologous cancer cell lines by direct recognition and antibody directed cellular cytotoxicity. J Exp Clin Cancer Res. 2010 Oct 11;29(1):134. doi: 10.1186/1756-9966-29-134. PMID 20937115